CLINICAL TRIAL: NCT01822210
Title: Botulinum Toxin (BOTOX) for Stomach Cancer Treatment
Brief Title: Botulinum Toxin for Stomach Cancer Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: StOlav2205; 2012-002493-31 (EudraCT Number)
Record Dates: First submitted 2013-03-21; First posted 2013-04-02 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Stomach Neoplasms
Keywords: Botulinum Toxins; Injections; Stomach; Tomography, X-Ray Computed
MeSH Terms: conditions — Stomach Neoplasms | interventions — Botulinum Toxins, Type A; Botulinum Toxins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Botox (Experimental): Injection of Botox in the tumor and surrounding stomach wall.
  Interventions: Drug: Botox

INTERVENTIONS:
Drug: Botox — injection by gastroscopy (100 Allergen units)
  Other Names: Botulinum toxin

SUMMARY:
Preclinical studies at our institution, using a genetic mouse model of gastric cancer, strongly suggest that innervation of the stomach wall is required not only for the development, but also for the progression of gastric cancer, and that denervation of the stomach either by vagotomy or by injection of botulinum toxin (Botox®) in the stomach wall may represent an effective therapeutic intervention. New treatment options for inoperable cancer in the stomach are urgently needed, and local treatment with botulinum toxin seems to be an attractive possibility. In this pilot study Botox injections will be given by gastroscopy in both the tumor and the surrounding stomach wall. The purpose of the study is to obtain data needed to calculate sample size in a larger controlled trial.

ELIGIBILITY:
Inclusion criteria:

Patients with verified gastric adenocarcinoma but found non-resectable or inoperable after evaluation in the appropriate multidisciplinary team at St.Olav Hospital. Trondheim University Hospital. The inclusion criteria for such patients are:

1. Patients who have received 1.line and 2. line chemotherapy but no longer respond to such therapy.
2. Patients who, due to toxicity of chemotherapy, cannot be offered such treatment.
3. Patients who, after meticulous information about chemotherapy, still do not want such treatment.
4. Patients with performance status (ECOG) 0-2.

Exclusion criteria:

1. Known allergy to any of the components in Botox®
2. Known peripheral motor neuropathy disease ( for example: Amyotrophic Lateral Sclerosis, ALS), or subclinical or clinical deficiency of neuromuscular transmission (for example: Myasthenia Gravis or Eaton-Lambert's Syndrome).
3. Pregnant or lactating women.
4. Another cancer disease that is not under control.
5. Another concomitant treatment for cancer.
6. Serious mental illness.
7. Performance status (ECOG) 3-4.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change of tumor volume in the stomach. | Baseline and 8 weeks
  Change measured with a standardized CT protocol (Thickness of the stomach wall and diameter of the tumor).
Change of tumor volume in the stomach. | 8 weeks and 20 weeks
  Change measured with a standardized CT protocol (Thickness of the stomach wall and diameter of the tumor).

SECONDARY OUTCOMES:
Toxicity | 2 weeks
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Toxicity | 8 weeks
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
performance status | 2 weeks
  ECOG scale
performance status | 8 weeks
  ECOG scale
performance status | 20 weeks
  ECOG scale

CONTACTS AND LOCATIONS:
Overall Officials: Jon Erik Grønbech, MD. PhD., Principal Investigator — St. Olavs Hospital
Locations (1):
- Department of Gastrointestinal Surgery, St Olavs Hospital Trondheim University Hospital, Trondheim, Norway

REFERENCES:
- [Result] Andersen G, Zhao CM, Cai X, Rabben HL, Fox JG, Wang TC, Chen D, Gronbech JE. Tu1418 Intragastric Injection of Botulinum Toxin a to Treat Gastric Cancer: An Open-Label Phase II Clinical Trial. Gastroenterology 150: S1251-1252, 2016 https://doi.org/10.1016/S0016-5085(16)34227-5